CLINICAL TRIAL: NCT07264556
Title: Effect of Opioid-Free, Opioid-sparing Versus Opioid-based Anesthesia on Perioperative NETs and Cancer Cell Malignancy in Patients Undergoing Surgery for Colorectal Cancer: A Randomized, Controlled Trial
Brief Title: Effect of OFA, OSA Versus Opioid-based Anesthesia on NETs and Cancer Cell Malignancy After Colorectal Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jun Zhang, Director, Head of Department of Anesthesiology,Principal Investigator, Clinical Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: OFA in CRC patients
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer; Opioid-free Anesthesia; NETs
Keywords: Opioid free anesthesia; Neutrophil extracellular trapping markers; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OA group (Experimental): petients received opioid-based anesthesia
  Interventions: Other: OA strategy
- OSA group (Experimental): patients received opioid-sparing anesthesia
  Interventions: Other: OSA stategy
- OFA group (Experimental): patients received opioid-free anesthesia
  Interventions: Other: OFA strategy

INTERVENTIONS:
Other: OA strategy — For OA group, anesthesia induction was conducted with an intravenous targeted control infusion (TCI) of 3-4 μg/mL propofol (effect-site concentration, Marsh mode), 2-3 ng/mL remifentanil (effect-site concentration, Minto mode), 0.5 μg/kg sufentanil, and 0.6 mg/kg rocuronium. General anesthesia was maintained with a continuous TCI infusion of 3 to 4 μg/mL propofol and 1 to 2 ng/mL remifentanil, intermittently administrated sufentanil and rocuronium. Patient controlled intravenous analgesia (PCIA) was performed with 0.5μg/ml of sufentanil and 0.75 mg/mL flurbiprofen after surgery. The PCIA scheme was set with the continuous infusion rate of 4 ml/h and single bolus injection volume of 4ml. The locking time was 15 min, and the PCIA was stopped 48 h after surgery.
  Arms: OA group
Other: OSA stategy — For OSA group, anesthesia induction was conducted with an intravenous targeted control infusion (TCI) of 3 to 4 μg/mL propofol, 2 to 3 ng/mL remifentanil, 0.3 μg/kg sufentanil, and 0.6 mg/kg rocuronium. After intubation, the patient received ultrasound-guided transversus abdominis plane (TAP) nerve block, with 0.375% ropivacaine 40mL injection. General anesthesia maintenance was consistent with OA group. Patient controlled intravenous analgesia (PCIA) was performed with 1mg/mL of oxycodone and 0.75 mg/mL flurbiprofen after surgery. The PCIA scheme was set with the continuous infusion rate was 4 ml/h and single bolus injection of 4ml. The locking time was 15 min, and the PCIA was stopped 48 hours after surgery.
  Arms: OSA group
Other: OFA strategy — For OFA group, before induction, an epidural catheter was inserted , and the catheter was advanced 4 cm cephalad. When the aspiration test results for blood and cerebrospinal fluid were negative, a test dose of lidocaine 1% (3 ml) was injected through the catheter. Ropivacaine (0.25%) was maintained at a rate of 5 ml/h during surgery. Anesthesia induction was conducted with an intravenous targeted control infusion (TCI) of 3-4 μg/mL propofol, 0.6 mg/kg rocuronium, 0.5mg/kg esketamine, 1mg/kg lidocaine and 0.5ug/kg dexmedetomidine. General anesthesia was maintained with a continuous TCI infusion of 3 to 4 μg/mL propofol, 1.5-mg/kg/h continuous infusion of lidocaine, 0.25 mg/kg/h continuous infusion of esketamine. At the postoperative stage, the epidural administration regimen included 0.15% ropivacaine. The continuous infusion rate was 5ml/h, with an additional 5 ml upon the patient's request, and the locking time was 15 min. The epidural catheter was removed 48 hours after surgery.
  Arms: OFA group

SUMMARY:
Adult patients aged 18-80 years old, American Society of Anesthesiologists physical status I-III, who were scheduled for elective colorectal cancer surgery under general anesthesia were recruited for this study. They were randomized to receive opioid-free anesthesia (OFA), opioid-sparing anesthesia (OSA) and opioid-based anesthesia (OA) group.

Blood samples were collected pre-surgery and 24h post-surgery. As primary endpoint, serum neutrophil myeloperoxidase (MPO) and citrullinated histone3 (CitH3) was measured. The secondary endpoints included the effects of postoperative serum on colorectal cancer (CRC) cells malignancy, numerical rating scale (NRS) scores, postoperative adverse events and recovery profiles.

For OA group, intraoperative remifentanil and sufentanil were used and postoperative patient controlled intravenous analgesia (PCIA) was performed with 0.5μg/ml of sufentanil and 0.75 mg/mL flurbiprofen, and the PCIA was stopped 48 h after surgery.

For OSA group, remifentanil and sufentanil were used only for anesthetic induction and the patient received ultrasound-guided transversus abdominis plane (TAP) nerve blockwas performed. Patient controlled intravenous analgesia (PCIA) was performed with 1mg/mL of oxycodone and 0.75 mg/mL flurbiprofen after surgery, and the PCIA was stopped 48 hours after surgery.

For OFA group, intraoperative epidural anesthesia combined with general anesthesia was used, and esketamine, lidocaine and dexmedetomidine for analgesia. Patient controlled epidural analgesia (PCEA) was used and terminated 48 hours after surgery.

DETAILED DESCRIPTION:
Adult patients aged 18-80 years old, American Society of Anesthesiologists physical status I-III, who were scheduled for elective colorectal cancer surgery under general anesthesia with endotracheal tube were recruited for this study. Tthey were randomized to receive opioid-free anesthesia (OFA), opioid-sparing anesthesia (OSA) and opioid-based anesthesia (OA) group.Blood samples were collected pre-surgery and 24h post-surgery. As primary endpoint, serum neutrophil myeloperoxidase (MPO) was detected. The secondary endpoints included the effects of postoperative serum on colorectal cancer (CRC) cells malignancy, numerical rating scale (NRS) scores, side effects and postoperative complications.

For OA group, anesthesia induction was conducted with an intravenous targeted control infusion (TCI) of 3-4 μg/mL propofol (effect-site concentration, Marsh mode), 2-3 ng/mL remifentanil (effect-site concentration, Minto mode), 0.5 μg/kg sufentanil, and 0.6 mg/kg rocuronium. General anesthesia was maintained with a continuous TCI infusion of 3 to 4 μg/mL propofol and 1 to 2 ng/mL remifentanil, intermittently administrated sufentanil and rocuronium. Patient controlled intravenous analgesia (PCIA) was performed with 0.5μg/ml of sufentanil and 0.75 mg/mL flurbiprofen after surgery. The PCIA scheme was set with the continuous infusion rate of 4 ml/h and single bolus injection volume of 4ml. The locking time was 15 min, and the PCIA was stopped 48 h after surgery.

For OSA group, anesthesia induction was conducted with an intravenous targeted control infusion (TCI) of 3 to 4 μg/mL propofol, 2 to 3 ng/mL remifentanil, 0.3 μg/kg sufentanil, and 0.6 mg/kg rocuronium. After intubation, the patient received ultrasound-guided transversus abdominis plane (TAP) nerve block, with 0.375% ropivacaine 40mL injection. General anesthesia maintenance was consistent with OA group. Patient controlled intravenous analgesia (PCIA) was performed with 1mg/mL of oxycodone and 0.75 mg/mL flurbiprofen after surgery. The PCIA scheme was set with the continuous infusion rate was 4 ml/h and single bolus injection of 4ml. The locking time was 15 min, and the PCIA was stopped 48 hours after surgery.

For OFA group, before induction, an epidural catheter was inserted under sterile conditions using the "loss-of-resistance" technique, and the catheter was advanced 4 cm cephalad. When the aspiration test results for blood and cerebrospinal fluid were negative, a test dose of lidocaine 1% (3 ml) was injected through the catheter. Ropivacaine (0.25%) was maintained at a rate of 5 ml/h during surgery. Anesthesia induction was conducted with an intravenous targeted control infusion (TCI) of 3-4 μg/mL propofol, 0.6 mg/kg rocuronium, 0.5mg/kg esketamine, 1mg/kg lidocaine and 0.5ug/kg dexmedetomidine. General anesthesia was maintained with a continuous TCI infusion of 3 to 4 μg/mL propofol, 1.5-mg/kg/h continuous infusion of lidocaine, 0.25 mg/kg/h continuous infusion of esketamine. At the postoperative stage, the epidural administration regimen included 0.15% ropivacaine. The continuous infusion rate was 5ml/h, with an additional 5 ml upon the patient's request, and the locking time was 15 min. The epidural catheter was removed 48 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-80 years old,
* American Society of Anesthesiologists physical status I-III,
* elective colorectal cancer surgery under general anesthesia

Exclusion Criteria:

* previous history of colorectal surgery,
* addicted to opioids,
* serious major mental or physical illness (heart, pulmonary, hepatic, or renal diseases),
* radiotherapy or chemotherapy history within 8 weeks prior to the surgery,
* contraindications to anesthetic agents or epidural.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
serum NETs biomarkers levels . | Day 1 before surgery and day 1 after surgery
  serum levels of neutrophil myeloperoxidase (MPO) and citrullinated histone3 (CitH3)

SECONDARY OUTCOMES:
colorectal cancer (CRC) cells malignancy | Day 1 after surgery
  the effects of postoperative serum on CRC cells proliferation, migration and invasion
numerical rating scale (NRS) scorespain score | Day 1 and day 2 after surgery
  numerical rating scale (NRS) scores at rest and on cough,NRS score is a scale of 0 to 10, the higher the score, the greater the degree of pain.
adverse event: postoperative nausea and vomiting | Day 1 and day 2 after surgery
  The incidence of the postoperative nausea and vomiting, ask the patient bedside if they have any complaints of nausea or vomiting postoperatively.
postoperative complications | On the day of surgery to the day discharge from hospital
  surgical complications
postoperative rcovery profiles | On the day of surgery to the day discharge from hospital
  length of PACU and hospital stay
postoperative rcovery profiles | Day 1 and day 2 after surgery
  first postoperative flatus,was defined as the proportion of patients passage of flatus or stool within 24 and 48 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No